CLINICAL TRIAL: NCT02460575
Title: L. Reuteri for Pediatric Diarrhea in Peru: Growth, Enteropathy, and Microbiota
Brief Title: Safety of Lactobacillus Reuteri in Healthy Children Aged 2-24 Months
Acronym: PRIDEC Peru
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tulane University School of Medicine (Other)
Collaborators: Johns Hopkins Bloomberg School of Public Health (Other); Asociacion Benefica Prisma (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); University of Virginia (Other)
Responsible Party: Principal Investigator, Richard A. Oberhelman, Professor, Tulane University School of Medicine
Organization: Tulane University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: U01DK105849 (NIH); U01DK105849 (NIH)
Record Dates: First submitted 2015-05-28; First posted 2015-06-02 (Estimated); Results first posted 2020-05-04 (Actual); Last update posted 2020-05-04 (Actual); Status verified 2020-04

CONDITIONS: Healthy
Keywords: Safety

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lactobacillus (Experimental): Active Product: Description Lactobacillus reuteri 17938 suspended in sunflower oil, medium chain triglyceride oil, silicone dioxide. Total viable count of L. reuteri 17938 1 x 108 CFU/5 drops.
  Interventions: Biological: Lactobacillus reuteri 17938
- Placebo (Placebo Comparator): Composition Sunflower oil, medium chain triglyceride oil and silicon dioxide. Total viable count of L. reuteri is zero CFU/ 5 drops.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Lactobacillus reuteri 17938 — probiotic
  Arms: Lactobacillus
Biological: Placebo — Composition Sunflower oil, medium chain triglyceride oil and silicon dioxide. Total viable count of L. reuteri is zero CFU/ 5 drops.
  Arms: Placebo

SUMMARY:
Phase I double blinded randomized trial of the safety and tolerability of Lactobacillus reuteri DSM 17938 given for five successive days in healthy children. Sixty children will receive study product at a treatment to placebo ratio of 2:1 and followed for 3 months for safety outcomes.

DETAILED DESCRIPTION:
The study is a single center Phase 1 double blind placebo controlled trial of Lactobacillus reuteri DSM 17938 in children aged 2-24 months. The study population is based in a community with a registered clinical trial center in rural Peru where this protocol can be done in a highly controlled setting. The study is intended to enroll healthy children living in a resource constrained setting where chronic undernutrition and diarrheal disease is common, as this is the population that is most likely to receive benefit from the use of this and or other probiotic products for the treatment of acute infectious diarrhea and environmental enteropathy.

Up to 100 subjects will be enrolled in order to obtain the randomization of 60 subjects, who will receive study product or placebo at a ratio of 2:1. Participants will be enrolled between the ages of 8 weeks and 24 months. There will be no age stratification. Participants will be screened with a baseline history and physical examination and laboratory tests to determine the HIV status of the child, as well baseline laboratory tests to evaluate occult infections, hepatic function, and renal function. Upon randomization subjects will be screened and randomized to a treatment arm. Product will be administered under the direct supervision of study staff daily for 5 days. The primary outcome is the safety and tolerability of the product at this dose and formulation. Safety will be assessed by the monitoring of baseline laboratory tests at 5 and 28 days following the initiation of therapy and by AE monitoring. Tolerability will be evaluated by analyzing 28 day diary cards that are distributed to all randomized subjects on which parents record their child's symptoms (specifically fever, anorexia/oral intake, vomiting, diarrhea, irritability, rash, wheezing, or open fields which allows them to describe any issue their child may experience and grade its severity) . Secondary outcomes include:

1) The assessment of the duration of shedding of Lactobacillus reuteri (Lr) strain DSM 17938 following administration. This will be determined by and endpoint PCR assay for L. reuteri done on stool collected on D3, D5, D12, D15, D18, D24, D28, D36 on all participants.

The planned enrollment period is four months and the participation of individual subjects is for 3 months. The study should be completed in 7 months. Safety monitoring by treatment group, i.e., infants assigned to active or placebo study product will be conducted by NIDDK appointed DSMB under the direction of the NIDDK Program Official.

ELIGIBILITY:
Inclusion Criteria:

* In order to be eligible to participate in this study, a subject must meet all of the following criteria:

  * Have a parental permission form signed by both parents
  * Be between 8 weeks to 24 months of age with no preexisting exclusion criteria
  * Have parents who are willing to comply with all planned study procedures and be available for planned study visits for 3 months.

Exclusion Criteria:

* 1) No enrollment of family members in households where any of the following are present:

  1. Another study participant in the household
  2. Presence of immune suppressed individuals or use of immunosuppressive agents (including but not limited to corticosteroids, methotrexate, etc.) by any household member
  3. Presence of a serious congenital anomaly or chronic medical condition that in the opinion of the investigators would contraindicate participation in any household member, including history of gastrointestinal surgery, chronic gastrointestinal illness, abnormal intestinal anatomy, or abnormal bowel functionality

     The following risk factors are at the level of the individual child:

     2) Allergy to penicillin, cephalosporins, clindamycin or gentamicin 3) History of antibiotic use in the last 30 days 4) Use of probiotic products within the past 30 days, including masato (local product with fermenting bacteria) and yogurt products containing live bacterial cultures.

     5) History of diarrheal illness within the past 30 days (See definition in Protocol Appendix B) 6) Presence of fever or a pre-existing adverse event monitored in the study (See Protocol Appendix B Definitions of AEs for specific adverse events monitored in the study) 7) Positive results on serum diagnostic tests for antibodies to HIV.

     8) Presence of severe anemia, defined as serum hemoglobin < 7 gm/dL

     9) Out of range laboratory values for total leucocyte count, BUN, Creatinine, AST, ALT, and total bilirubin monitored as potential adverse events, as described in Appendix E.

     10) Pre-enrollment stool sample (collected within 14 days of day 1 of the study) is positive for L. reuteri by PCR.

Ages: 2 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2019-01-09 (Actual); Primary Completion 2019-12-29 (Actual); Study Completion 2019-12-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret N Kosek, MD, Principal Investigator — University of Virginia
Locations (1):
- Centro de Salud de Santa Clara, Santa Clara, Loreto, Peru

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lactobacillus | Placebo
Started | 40 | 20
Completed | 39 | 20
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lactobacillus | Placebo | Total
Number analyzed (Participants) | 40 | 20 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 40 | 20 | 60
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: months] | 10.5 (5.8) | 11.9 (5.2) | 10.9 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 12 | 29
  Male | 23 | 8 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 40 | 20 | 60
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Peru | 40 | 20 | 60

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Positive Blood Culture for L. Reuteri
Description: number of participants with positive blood culture for L. reuteri
Time Frame: Participants are followed for an average of 36 days
Measure: Count of Participants; unit: Participants
Arm/Group | Lactobacillus | Placebo
Number analyzed (Participants) | 40 | 20
Participants | 0 | 0

2. Primary Outcome: Mean Daily Temperature
Time Frame: 5 days of study product administration
Measure: Mean (Standard Deviation); unit: degrees Centigrade/day
Arm/Group | Lactobacillus | Placebo
Number analyzed (Participants) | 40 | 20
degrees Centigrade/day | 36.5 (0.23) | 36.5 (0.23)

ADVERSE EVENTS:
Time Frame: 3 month followup period
Description: same as clinicaltrials.gov definition
Arm/Group | Lactobacillus | Placebo
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/20
Other Adverse Events (participants affected / at risk) | 28/40 | 16/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lactobacillus (N=40) | Placebo (N=20)
All (General disorders) | 28 (43) | 16 (27) — All non serious AEs
Fever (General disorders) | 17 (17) | 9 (9)
Diarrhea (Gastrointestinal disorders) | 13 (13) | 7 (7)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1)
Irritability (General disorders) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Pruritis (General disorders) | 1 (1) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Informed Consent Form (2017-08-11): https://cdn.clinicaltrials.gov/large-docs/75/NCT02460575/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2019-01-11): https://cdn.clinicaltrials.gov/large-docs/75/NCT02460575/Prot_SAP_001.pdf